CLINICAL TRIAL: NCT02420691
Title: A Phase II Study of LEE011 (Ribociclib) in Patients With Advanced Neuroendocrine Tumors of Foregut Origin
Brief Title: Ribociclib in Treating Patients With Advanced Neuroendocrine Tumors of Foregut Origin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0371; NCI-2015-01017 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0371 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Advanced Digestive System Neuroendocrine Neoplasm; Duodenal Neuroendocrine Tumor G1; Functional Pancreatic Neuroendocrine Tumor; Gastric Neuroendocrine Tumor; Intermediate Grade Lung Neuroendocrine Neoplasm; Low Grade Lung Neuroendocrine Neoplasm; Nonfunctional Pancreatic Neuroendocrine Tumor; Thymus Neoplasm
MeSH Terms: conditions — Non functioning pancreatic endocrine tumor; Thymus Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ribociclib) (Experimental): Patients receive ribociclib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ribociclib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011

SUMMARY:
This phase II trial studies how well ribociclib works in treating patients with neuroendocrine tumors of the foregut, which includes the thymus, lung, stomach, and pancreas, that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced tumors). Ribociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the Response Evaluation Criteria in Solid Tumors (RECIST) (per version 1.1) objective response rate of LEE011 (ribociclib) among patients with advanced foregut neuroendocrine tumors (NETs).

SECONDARY OBJECTIVES:

I. To evaluate the progression free survival duration of LEE011 among patients with advanced foregut NETs.

II. To evaluate the safety and tolerability of LEE011 in patients with advanced foregut NETs.

III. To determine clinic benefit rate at 6 months (defined as complete response plus partial response plus stable disease) with LEE011 among patients with advanced foregut NETs.

EXPLORATORY OBJECTIVES:

I. To determine baseline molecular markers (mutations, deletions, and amplifications in multiple endocrine neoplasia [MEN]1, p27, p16 and cyclin D1 [CCND1]) in archival tumor that may predict clinical benefit at 6 months from LEE011.

II. To determine potential mechanisms/markers of resistance. III. To determine early chromogranin and neuron specific enolase responses in patients with elevated levels at baseline.

IV. To determine the pharmacodynamic changes including proliferation-related Ki-67 antigen (Ki-67) and phosphorylated retinoblastoma (pRb) upon treatment with LEE011 in patients with advanced foregut NETs.

OUTLINE:

Patients receive ribociclib orally (PO) once daily (QD) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed low or intermediate grade, unresectable well differentiated foregut neuroendocrine tumors (thymic, bronchopulmonary, gastric, duodenal and pancreatic); patients with multiple neuroendocrine tumors associated with MEN1 syndrome will be eligible
* Patients must have radiographically measurable disease
* Pancreatic neuroendocrine patients must have had progression after prior therapy; patients with other foregut neuroendocrine tumors must have had progressive disease over the last 12 months, irrespective of prior therapy; patients with both functional (who may continue somatostatin analogues as required for control of related symptoms) and non-functional tumors are eligible; in patients who have previously received therapy, the number of prior lines of therapy should not be more than 2 lines of systemic therapy not including somatostatin analogues
* Written informed consent must be obtained prior to any screening procedures
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* A sufficient interval must have elapsed between the last dose of prior anti-cancer therapy (including cytotoxic and biological therapies and major surgery) and enrollment, to allow the effects of prior therapy to have abated: a) cytotoxic or targeted chemotherapy: greater than or equal to the duration of the cycle of the most recent treatment regimen (a minimum of 3 weeks for all regimens, except 6 weeks for nitrosoureas and mitomycin-C); b) biologic therapy (e.g., antibodies): greater than or equal to 4 weeks
* Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L
* Hemoglobin (Hgb) greater than or equal to 9 g/dL
* Platelets greater than or equal to 100 x 10^9/L
* Serum total bilirubin less than or equal to 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) less than or equal to 2.5 x ULN, except in patients with tumor involvement of the liver who must have AST and ALT less than or equal to 5 x ULN
* Serum creatinine less than or equal to 1.5 x ULN or 24-hour clearance greater than or equal to 50 mL/min
* Serum potassium (corrected for serum albumin) must be within clinically relevant limits (e.g., a patient can be enrolled if a lab value may be outside the normal laboratory range but the abnormality is not clinically relevant or can be repleted)
* Sodium (corrected for serum albumin) must be within clinically relevant limits (e.g., a patient can be enrolled if a lab value may be outside the normal laboratory range but the abnormality is not clinically relevant or can be repleted)
* Magnesium (corrected for serum albumin) must be within clinically relevant limits (e.g., a patient can be enrolled if a lab value may be outside the normal laboratory range but the abnormality is not clinically relevant or can be repleted)
* Phosphorus (corrected for serum albumin) must be within clinically relevant limits (e.g., a patient can be enrolled if a lab value may be outside the normal laboratory range but the abnormality is not clinically relevant or can be repleted)
* Total calcium (corrected for serum albumin) must be within clinically relevant limits (e.g., a patient can be enrolled if a lab value may be outside the normal laboratory range but the abnormality is not clinically relevant or can be repleted)
* Negative pregnancy test (serum beta-human chorionic gonadotropin [B-HCG]) within 7 days of starting study treatment is required in women of childbearing potential; NET patients with positive B-HCG are eligible if pregnancy can be excluded by vaginal ultrasound or lack of expected doubling of B-HCG

Exclusion Criteria:

* Patient has a known hypersensitivity to LEE011 or any of its excipients
* Patients with known or suspected brain metastases; however, if radiation therapy and/or surgery has been completed and serial evaluation by computed tomography (CT) (with contrast enhancement) or magnetic resonance imaging (MRI) over a minimum of 3 months demonstrates the disease to be stable and if the patient remains asymptomatic, then the patient may be enrolled; such patients must have no need for treatment with steroids or anti-epileptic medications
* Patients with concurrent malignancies or malignancies within 3 years prior to starting study drug (with the exception of tumors common to a single genetic cancer syndrome, i.e. MEN1, MEN2, von Hippel-Lindau [vHL], tuberous sclerosis complex [TSC] etc., or adequately treated, basal cell skin cancer, squamous cell carcinoma, non-melanoma skin cancer or curatively resected cervical cancer)
* Patient is not able to swallow oral medication and/or has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Known diagnosis of human immunodeficiency virus (HIV) or hepatitis C (testing is not mandatory)
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in the clinical study (e.g. chronic pancreatitis, chronic active hepatitis, etc.)
* Patient who has received radiotherapy within less than or equal to 4 weeks or limited field radiation for palliation within less than or equal to 2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom greater than or equal to 30% of the bone marrow was irradiated
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery)
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following: a) history of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis less than 12 months prior to screening b) history of documented congestive heart failure (New York Heart Association functional classification III-IV) c) documented cardiomyopathy d) patient has a left ventricular ejection fraction (LVEF) less than 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening e) history of ventricular, supraventricular, nodal arrhythmias, or any other cardiac arrhythmias, long QT syndrome or conduction abnormality within 12 months prior to starting study drug f) congenital long QT syndrome or a family history of corrected QT interval (QTc) prolongation g) on screening, inability to determine the corrected QT for Fridericia (QTcF) interval on the electrocardiogram (ECG) (i.e.: unreadable or not interpretable) or QTcF > 450 msec (using Fridericia's correction); all as determined by screening ECG (mean of triplicate ECGs)
* Systolic blood pressure greater than 160 mmHg or less than 90 mmHg at screening
* Patients who are currently receiving treatment with agents that are known to cause QTc prolongation or inducing Torsade de Pointes in humans and are unable to discontinue or switch to an alternate medication
* Patients who are currently receiving treatment (within 5 days prior to starting study drug) with agents that are known strong inducers or inhibitors of cytochrome P450, family 3, subfamily A polypeptide 4 (CYP3A4)/cytochrome P450, family 3, subfamily A polypeptide 5 (5), or that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
* Patients with concurrent severe and/or uncontrolled concurrent medical conditions that could compromise participation in the study (e.g., uncontrolled diabetes mellitus defined by a glucose greater than 1.5 ULN in spite of adequate medical treatment, clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection)
* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (greater than 5 mIU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation; highly effective contraception methods include: total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception; female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment; male sterilization (at least 6 months prior to screening); for female patients on the study, the vasectomized male partner should be the sole partner for that patient; combination of any of the two following (a+b or a+c or b+c) a. use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception b. placement of an intrauterine device (IUD) or intrauterine system (IUS) c. barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository; in case of use of oral contraception, women should have been stable on the same pill before taking study treatment; note: oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception; women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Sexually active males unless they use a condom during intercourse while taking the drug and for 21 days after stopping treatment and should not father a child in this period; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
* Patients unwilling or unable to comply with the protocol
* Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise; therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nageshwara V Dasari, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2015-August 2016. All patients enrolled at MD Anderson.
Pre-assignment Details: 21 participants consented, 1 participant was not eligible due to screen failure.
Groups:
- Study Participants: LEE011 will be taken orally, once a day for 21 consecutive days followed by a 7 day planned break. LEE011 will be dosed on a flat dosing scale of 600 mg/day, irrespective of size and weight.
Period: Overall Study
Arm/Group | Study Participants
Started | 20
Completed | 14
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 57 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Rate Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years 10 months
Measure: Number; unit: participants
Arm/Group | Study Participants
Number analyzed (Participants) | 19
participants | 19

2. Secondary Outcome: Number of Participants With Clinical Benefit Rate
Description: Number of Participants that did not have progressive disease at 6 months.
Time Frame: At 6 months
Measure: Number; unit: participants
Arm/Group | Study Participants
Number analyzed (Participants) | 19
participants | 19

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the length of time during and after the treatment that a participant lives with the disease but it does not get worse.The Kaplan-Meier (KM) method will be used to estimate the PFS.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study Participants
Number analyzed (Participants) | 20
months | 10.44 [7.37 to 13.49]

4. Other Pre Specified Outcome: Change in pRB With Treatment
Description: Decrease in pRB as Measured by Immunohistochemistry (IHC) in Biopsies From Baseline and From cycle 2 day 1. H-scores were calculated as the sum of the products of the percentage of positive staining areas and the staining intensity (0, 1, 2 or 3), and ranged from 0 to 300. A score of 0 represents the absence of expression, and an H-score of 300 represents maximum expression.
Time Frame: Baseline (Pre-Treatment) and Cycle 2 Day 1, each Cycle is 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 19
score on a scale
  H- Score Pre-Treatment | 236.47 (67.25)
  H-Score Post-Treatment | 238.32 (39.56)

5. Other Pre Specified Outcome: Change in Ki-67 With Treatment
Description: Ki-67 was calculated as a percentage cells staining positive by Immunohistochemistry (IHC).
Time Frame: Baseline (Pre-Treatment) and Cycle 2 Day 1, each Cycle is 28 days
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Study Participants
Number analyzed (Participants) | 19
percentage of cells
  Pre-Treatment | 13.61 (10.18)
  Post-Treatment | 19.11 (17.83)

ADVERSE EVENTS:
Time Frame: 3 years and 5 months
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 11/20
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Participants (N=20)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 2
Pneumothroax (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiac Chest Pain (General disorders) | 1
Encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Participants (N=20)
Neutrophil Count Increased (Investigations) | 17
Nausea (Metabolism and nutrition disorders) | 12
Anemia (Blood and lymphatic system disorders) | 12
Fatigue (General disorders) | 11
Platelet Count Decreased (Investigations) | 9
Creatinine Increased (Investigations) | 8
Vomiting (Gastrointestinal disorders) | 5
Alanine Aminotransferase Increased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Aspartate Aminotransferase Increased (Investigations) | 3
Weight Loss (Investigations) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 3
Edema Limbs (General disorders) | 3
Dysguesia (Nervous system disorders) | 3
Fever (General disorders) | 2
Alkaline Phosphatase Increased (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Blood Bilirubin Increased (Investigations) | 2
Headache (Nervous system disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Urinary Tract Infection (Infections and infestations) | 1
Investigations: Other- Hyperphosphatemia (Investigations) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Skin infection (Infections and infestations) | 1
Malaise (General disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Edema Face (General disorders) | 1
Hematoma (Vascular disorders) | 1
Abdominal Distention (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Eye Disorders: Other- Periorbital Swelling and Crystal Discharge (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02420691/Prot_SAP_000.pdf